CLINICAL TRIAL: NCT01200784
Title: Dose Finding Study of Nicotinamide in Hemodialysis Patients With Hyperphosphatemia
Brief Title: Nicotinamide in Hemodialysis Patients With Hyperphosphatemia
Acronym: DONATO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medice Arzneimittel Pütter GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6520-9961-03; 2009-015821-34 (EudraCT Number)
Record Dates: First submitted 2010-09-10; First posted 2010-09-14 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Kidney Disease; Hemodialysis; Hyperphosphatemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 250 mg/d modified release Nicotinamide (Experimental)
  Interventions: Drug: Nicotinamide
- 500 mg/d modified release Nicotinamide (Experimental)
  Interventions: Drug: Nicotinamide
- 750 mg/d modified release Nicotinamide (Experimental)
  Interventions: Drug: Nicotinamide
- 1000 mg/d modified release Nicotinamide (Experimental)
  Interventions: Drug: Nicotinamide
- 1000 mg/d immidiate release Nicotinamide (Active Comparator)
  Interventions: Drug: Nicotinamide

INTERVENTIONS:
Drug: Nicotinamide — dosage

SUMMARY:
Study hypothesis: Nicotinamide inhibits gastrointestinal phosphate absorption and serum phosphate levels of dialysis patients in a dose dependent manner.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis since 3 months or longer
* hemodialysis frequency 3 times weekly
* stable phosphate binder dose since one month at screening
* serum phosphate level < 2,42 mmol/l at screening
* serum phosphate level > 1,52 mmol/l after wash out phase
* stable treatment with vitamin D analogues since one month at screening

Exclusion Criteria:

* congestive heart failure
* acute bleeding complications
* acute myocardial infarction
* peptic ulcers
* serious liver damage
* poorly controlled diabetes
* severe visual impairment
* uncontrolled high blood pressure
* thrombocyte count < 120/nl
* difficulties in swallowing or dysphagia
* diminished intestinal motility, megacolon, pseudo- or mechanical obstruction
* gastroparesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
serum phosphate | 4 weeks of active treatment

SECONDARY OUTCOMES:
serum phosphate | 8 weeks of active treatment
serum calcium | 4 and 8 weeks of acitve treatment
serum PTH | 4 and 8 weeks of active treatment
adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Walter Zidek, Prof. Dr., Study Director — Charité Berlin, Campus Benjamin Franklin, Innere Medizinische Klinik IV WE 28
Locations (33):
- Germany (33):
  - Alsfeld
  - Arnstadt
  - Augsburg
  - Berlin
  - Bielefeld
  - Coburg
  - Darmstadt
  - Dortmund
  - Dülmen
  - Düsseldorf
  - Elsenfeld
  - Erfurt
  - Essen
  - Friedrichsroda
  - Hamburg
  - Hamelin
  - Hellersdorf
  - Herne
  - Herzberg
  - Iserlohn
  - Jena-Drakendorf
  - Kamen
  - Kreuzberg
  - Leverkusen
  - Mannheim
  - Minden
  - Nordhausen
  - Osnabrück
  - Pfarrkirchen
  - Regensburg
  - Schwabach
  - Tangermünde
  - Wuppertal